CLINICAL TRIAL: NCT05836935
Title: Role of Imaging in Complications of Sinusitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Mohamed, Resident of radiology at sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-04-02MS
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Rhinosinusitis; Intracranial Extension; Rhinosinusitis Chronic; Rhinosinusitis Acute; Fungal Sinusitis; Allergic Fungal Rhinosinusitis; Invasive Fungal Sinusitis (Diagnosis)
Keywords: Rhinosinusitis; complicated sinusitis; complications of sinusitis; Magnetic resonance imaging; Computed tompgraphy; MRI; CT
MeSH Terms: conditions — Rhinosinusitis; Allergic Fungal Sinusitis; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental)
  Interventions: Radiation: Multislice CT scan of the paranasal sinuses.; Radiation: MRI examination of the paranasal sinuses

INTERVENTIONS:
Radiation: Multislice CT scan of the paranasal sinuses. — MSCT scan using GE Revolution Evo 128 multidetector elements scanner (GE Healthcare, Chicago, Illinois, United state) , Toshiba Alexion 16 detector elements scanner (Aplio 500, Toshiba Medical Systems, Otawara-shi, Tochigi 324-8550, Japan). Or Canon Aquilion Prime SP 160 -multidetector- row CT scanner (Canon Medical Systems, Tochigi, Japan) Thin slice Axial scans will be taken at 0.625-1.0 mm slice thickness, commencing from the hard palate till above the end of frontal sinuses, coronal and sagittal multiplanar reconstruction images will be obtained.
Radiation: MRI examination of the paranasal sinuses — MRI imaging using Philips Achieva 1.5T MRI device (Philips Achieva, Netherlands) or Siemens Magnetom Altea 1.5T MRI device (Siemens Healthineers, Germany) for suspected intracranial and orbital complications.

SUMMARY:
This study aims to assess the diagnostic performance of CT and MRI in the diagnosis of complications of rhinosinusitis in comparison to clinical and operative findings.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed as sinusitis with clinically suspected complications through history and physical examination (site, onset, character of pain, constitutional symptoms, duration).

Exclusion Criteria:

* Patients with absolute or relative contraindications for cross sectional imaging including; claustrophobia, metallic implants, pacemaker and prosthetic heart valves for MRI.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of different Types of possible complications detected by CT and MRI | 6 months
  To diagnose the diagnostic accuracy of CT and MRI in detection of different types of orbital and intracranial complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carr TF. Complications of sinusitis. Am J Rhinol Allergy. 2016 Jul;30(4):241-5. doi: 10.2500/ajra.2016.30.4322. PMID 27456592
- [Background] Marchiano E, Raikundalia MD, Carniol ET, Echanique KA, Kalyoussef E, Baredes S, Eloy JA. Characteristics of patients treated for orbital cellulitis: An analysis of inpatient data. Laryngoscope. 2016 Mar;126(3):554-9. doi: 10.1002/lary.25529. Epub 2015 Aug 26. PMID 26307941
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Background] Chen CY, Sheng WH, Cheng A, Chen YC, Tsay W, Tang JL, Huang SY, Chang SC, Tien HF. Invasive fungal sinusitis in patients with hematological malignancy: 15 years experience in a single university hospital in Taiwan. BMC Infect Dis. 2011 Sep 22;11:250. doi: 10.1186/1471-2334-11-250. PMID 21939544
- [Background] Chakrabarti A, Denning DW, Ferguson BJ, Ponikau J, Buzina W, Kita H, Marple B, Panda N, Vlaminck S, Kauffmann-Lacroix C, Das A, Singh P, Taj-Aldeen SJ, Kantarcioglu AS, Handa KK, Gupta A, Thungabathra M, Shivaprakash MR, Bal A, Fothergill A, Radotra BD. Fungal rhinosinusitis: a categorization and definitional schema addressing current controversies. Laryngoscope. 2009 Sep;119(9):1809-18. doi: 10.1002/lary.20520. PMID 19544383